CLINICAL TRIAL: NCT06861283
Title: Development and Validation of a Digital Twin-based Clinical Research System (X Town Stage I)
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Collaborators: Tsinghua University (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Li Huating, Professor, Shanghai 6th People's Hospital
Other Study IDs: 2025-KY-025(K)
Record Dates: First submitted 2025-02-18; First posted 2025-03-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-02

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Virtual clinical studies
- Real-world clinical studies

SUMMARY:
Chronic diseases, characterized by their prolonged duration and slow progression, have emerged as predominant contributors to global morbidity and mortality. The investigators have developed a digital twin-based clinical research system (termed X Town) for chronic diseases, to predict clinical outcomes under various interventions. In this study, the investigators aim to evaluate the reliability of the developed digital twin-based clinical research system in predicting short-term clinical outcomes via virtual and real-world clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old
2. Receiving care at a community health service centre
3. Able to understand and comply with the study procedures
4. Agrees to participate in the study and signs the informed consent form

Exclusion Criteria:

1. Patients with severe mental illness
2. Patients expected to be unable to complete follow-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will mainly include participants at high-risk of or with chronic diseases.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-04-13 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
The agreement between the simulated short-term clinical outcomes in the virtual clinical studies and the real-world short-term clinical outcomes in the real-world clinical studies | Within 3 months
  We will use three predefined binary metrics to evaluate the agreement: (1) full statistical significance agreement, defined by effect estimates and CIs of the virtual and real-world clinical studies on the same side of the null; (2) estimate agreement, defined by whether effect estimates for the virtual clinical studies fell within the 95% CI for the real-world clinical study results; (3) standardized difference agreement between treatment effect estimates from the real-world clinical studies and the virtual clinical studies, defined by standardized differences (Reference: JAMA. 2023;329(16):1376-1385. doi:10.1001/jama.2023.4221).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Health and Medical Center, Wuxi, Jiangsu, China